CLINICAL TRIAL: NCT01738737
Title: Effect of Low-level Laser Therapy (904 nm) and Static Stretching in Patients With Knee Osteoarthritis: Randomised Controlled Trial.
Brief Title: Low-level Laser Therapy and Static Stretching in Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CAPPESQ 455/11
Record Dates: First submitted 2012-08-28; First posted 2012-11-30 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Stretching (Experimental): Seven stretching exercises for lower limbs during 24 sessions
  Interventions: Other: Stretching exercises
- Placebo laser + Stretching (Experimental): application of placebo laser therapy during nine sessions plus stretching exercises during 24 sessions
  Interventions: Other: Stretching exercises; Device: placebo laser therapy
- Active laser + Stretching (Experimental): application of active laser therapy during nine sessions plus stretching exercises during 24 sessions
  Interventions: Device: Active Laser; Other: Stretching exercises
- Active Laser (Experimental): Application of active laser only during 24 sessions
  Interventions: Device: Active Laser
- Control (No Intervention): Control group that will receive a small book with informations about knee osteoarthritis and postural orientation.

INTERVENTIONS:
Device: Active Laser — 18 points of application of active laser in the knee (frontal faces, lateral and medial)
  Other Names: LaserPulse (904nm) class II IBRAMED
  Arms: Active Laser; Active laser + Stretching
Other: Stretching exercises — 7 stretching exercises for lower limbs lasting 30 seconds with 4 repetitions
  Arms: Active laser + Stretching; Placebo laser + Stretching; Stretching
Device: placebo laser therapy — 18 points of application of placebo laser in the knee (frontal faces, lateral and medial)
  Other Names: LaserPulse class II IBRAMED
  Arms: Placebo laser + Stretching

SUMMARY:
Osteoarthritis (OA) is a highly prevalent and disabling disease. It is estimated that by 2030 the prevalence of symptomatic OA could reach 30% of the population above 60 years. It is associated with significant morbidity being one of the most common causes of joint pain, functional disability and compromised quality of life. This randomised controlled trial will investigate the effect of low-level laser therapy (LLLT) and static stretching exercises, as monotherapy and in combination, on pain, quality of life, function, mobility, knee range of motion (KROM) and hamstring length in participants with knee OA.

This study will involve 145 people aged 50-75 years with symptomatic radiographic knee OA and will consist of two types of treatments: Low-level laser therapy (LLLT) and stretching exercises. The patients will be randomly allocated to five study groups LLLT active+Stretch, LLLT placebo+Stretch, Stretch, LLLT and Control (with n=29 each). Treatment frequency will be three sessions/week for all active groups. LLLT will involve the use of a Galium-Arsenide laser (904nm, 40 milliwatts, 3 Joules/point, 27 Joules/knee) over 24 sessions for the monotherapy group and 9 sessions for the LLLT+Stretch groups. Stretching will consist of seven exercises completed over 24 sessions. The control group will receive a booklet.

The primary outcome is pain measured by Visual Analogue Scale. Secondary outcomes included quality of life assessed by Western Ontario and McMaster Universities Arthritis Index (WOMAC), function by Lequesne Algofunctional Index, mobility by Timed Up and Go Test (TUG), KROM by goniometry of knee flexion and hamstring shortening by popliteal angle. The statistical method will follow the principles of per-protocol analysis.

DETAILED DESCRIPTION:
Physical performance as a determinant of disability in osteoarthritis (OA) has been investigated extensively, but research has focused primarily on the effect that the decrease in muscle strength has on the functionality in patients with OA. However, the reduced range of motion in affected joints is also an important risk factor for the occurrence of locomotor disability and other developing disability in patients with OA.

Studies using stretching exercises are scarce in the Reid & Mc Nair (2010) specifically examined the range of motion can be improved in subjects with knee osteoarthritis, although this study did only stretching the hamstrings. The results indicate that there is immediate benefits of stretching in subjects with osteoarthritis of the knee joint, providing evidence for the long term development of stretching programs for this population.

In the literature are observed inconsistent results regarding the benefits of laser treatment in improving pain and function in individuals with knee OA. Also there are few studies that specify which dosage and frequency of laser must be used.

In view of the increasing need to support the role of physiotherapy in evidence-based practice, this study is justified by the need to test the effectiveness of stretching exercises and elucidate the effectiveness of low intensity laser therapy in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* radiographic evidence of knee osteoarthritis between 2-4 in Kellgren & Lawrence classification
* pain intensity ≥3 on a 10cm Visual Analogue Scale (VAS)
* knee symptoms for at least 3 months

Exclusion Criteria:

* symptomatic hip osteoarthritis
* any disease where laser treatment is contraindicated (cancer and uncontrolled diabetes mellitus)
* continuous use of anti-inflammatory drugs
* other concurrent injury/conditions that will affect their ability to participate in the rehabilitation program and/or assessment procedures.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rubia F Meneses, Principal Investigator — University of Sao Paulo
Locations (1):
- Specialized rehabilitation service, Taboão da Serra, São Paulo, Brazil

REFERENCES:
- [Derived] Ferreira de Meneses SR, Hunter DJ, Young Docko E, Pasqual Marques A. Effect of low-level laser therapy (904 nm) and static stretching in patients with knee osteoarthritis: a protocol of randomised controlled trial. BMC Musculoskelet Disord. 2015 Sep 14;16:252. doi: 10.1186/s12891-015-0709-9. PMID 26369333

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Laser + Stretching: application of placebo laser therapy during nine sessions plus stretching exercises during 24 sessions
  Stretching exercises: 7 stretching exercises for lower limbs lasting 30 seconds with 4 repetitions
  placebo laser therapy: 9 points of application of placebo laser per knee (frontal faces, lateral and medial)
- Active Laser + Stretching: application of active laser therapy during nine sessions plus stretching exercises during 24 sessions
  Active Laser: 9 points of application of active laser per knee (frontal faces, lateral and medial)
  Stretching exercises: 7 stretching exercises for lower limbs lasting 30 seconds with 4 repetitions
- Active Laser: Application of active laser only during 24 sessions
  Active Laser: 9 points of application of active laser per knee (frontal faces, lateral and medial)
Period: Overall Study
Arm/Group | Stretching | Placebo Laser + Stretching | Active Laser + Stretching | Active Laser | Control
Started | 29 | 29 | 29 | 29 | 29
Completed | 25 | 25 | 25 | 25 | 25
Not Completed | 4 | 4 | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Population: There was no statistically significant difference between groups at baseline (p> 0.05).
Groups:
- Total: Total of all reporting groups
Arm/Group | Stretching | Placebo Laser + Stretching | Active Laser + Stretching | Active Laser | Control | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.1) | 64.8 (6.3) | 62.7 (6.8) | 66.4 (5.9) | 62.4 (6.3) | 63.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 19 | 18 | 22 | 98
  Male | 8 | 3 | 6 | 7 | 3 | 27
Pain [Mean (Standard Deviation); unit: cm on Visual Analogue Scale (0-10)] — Scale varies from 0 (no pain) to 10 (worst pain possible).
  cm on Visual Analogue Scale (0-10) | 6.5 (1.4) | 6.5 (1.7) | 6.0 (2.2) | 5.7 (2.1) | 5.3 (1.9) | 6.0 (1.9)
Self-reported symptoms [Mean (Standard Deviation); unit: units on scale WOMAC] — Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) asses self reported symptoms of pain, function and stiffness. The total scores varies from 0 (no impairment) to 96 (worse outcome).
  units on scale WOMAC | 35.2 (14.8) | 33.4 (16.6) | 32.2 (14.8) | 39.5 (20.7) | 33.4 (17.6) | 34.7 (16.9)
Function [Mean (Standard Deviation); unit: units on Lequesne Functional Question.] — The questionnaire varies from 0 to 24. Higher values represent worse outcome.
  units on Lequesne Functional Question. | 10.1 (4.4) | 10.1 (4.7) | 10.7 (4.5) | 11.4 (5.6) | 9.3 (4.5) | 10.3 (4.7)
Mobility - Timed Get up and Go (TUG) [Mean (Standard Deviation); unit: seconds] — TUG measures the time a person spends to get up from a chair, walks at the usual speed for 3m, turns, walk back and sit down.
  seconds | 15.0 (3.0) | 15.8 (4.0) | 14.8 (4.0) | 16.0 (3.0) | 13.5 (2.4) | 15.0 (3.3)
Knee range of motion [Median (Inter-Quartile Range); unit: degrees] | 108.0 [93.5 to 115.2] | 106.0 [96.2 to 109.0] | 102.0 [88.0 to 116.0] | 93.0 [81.5 to 107.0] | 104.0 [100.7 to 112.7] | 102.6 [92.0 to 112.0]
Hamstring shortening [Median (Inter-Quartile Range); unit: degrees] | 20.0 [15.0 to 28.7] | 28.0 [20.7 to 32.5] | 25.0 [19.5 to 29.5] | 26.0 [15.0 to 39.0] | 24.0 [19.5 to 31.5] | 24.6 [17.9 to 32.2]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Analogue Scale for Pain
Description: The scale varies from 0 to 10. Higher values represent worse outcomes. The assessment will be done in the patient's first evaluation and after each intervention.
Time Frame: Baseline and post-intervention, up to 11 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Laser + Stretching | Placebo Laser + Stretching | Stretching | Active Laser | Control
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
units on a scale | 3.2 (2.1) | 3.8 (2.3) | 3.1 (2.9) | 3.3 (2.2) | 0.7 (3.0)

2. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index
Description: The scale varies from 0 to 96. Higher values represent worse outcomes. The assessment will be done in the patient's first evaluation and after each intervention.
Time Frame: Baseline and post-intervention, up to 11 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Laser + Stretching | Placebo Laser + Stretching | Stretching | Active Laser | Control
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
units on a scale | 8.0 [6.0 to 15.0] | 11.0 [4.5 to 21.5] | 13.0 [5.7 to 22.5] | 16.0 [8.7 to 24.5] | 2.0 [-2.5 to 8.5]

3. Secondary Outcome: Change From Baseline in Range of Motion of Flexion of the Knee
Description: Higher values represent better outcomes The assessment will be done in the patient's first evaluation and after each intervention.
Time Frame: Baseline and post-intervention, up to 11 weeks
Measure: Median (Inter-Quartile Range); unit: degress
Arm/Group | Active Laser + Stretching | Placebo Laser + Stretching | Stretching | Active Laser | Control
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
degress | 7.0 [3.0 to 15.0] | 10.0 [4.0 to 15.2] | 6.0 [-1.0 to 11.5] | 10.0 [-7.5 to 23.2] | 1.0 [-5.5 to 7.0]

4. Secondary Outcome: Change From Baseline in Lequesne Functional Questionnaire
Description: The scale varies from 0 to 24. Higher values represent worse outcomes The assessment will be done in the patient's first evaluation and after each intervention.
Time Frame: Baseline and post-intervention, up to 11 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Laser + Stretching | Placebo Laser + Stretching | Stretching | Active Laser | Control
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
units on a scale | 2.5 [0.4 to 5.1] | 1.5 [0.5 to 5.2] | 4.0 [0.5 to 6.6] | 3.5 [1.9 to 5.6] | 0.0 [-2.2 to 1.0]

5. Secondary Outcome: Change From Baseline in Timed Get Up and Go Test
Description: Higher values represent worse outcomes The assessment will be done in the patient's first evaluation and after each intervention.
Time Frame: Baseline and post-intervention, up to 11 weeks
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Active Laser + Stretching | Placebo Laser + Stretching | Stretching | Active Laser | Control
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
seconds | 2.5 [-0.2 to 4.7] | 3.0 [1.1 to 6.7] | 2.6 [1.3 to 4.1] | 3.1 [0.5 to 6.4] | 0.0 [-1.0 to 1.2]

ADVERSE EVENTS:
Arm/Group | Active Laser + Stretching | Placebo Laser + Stretching | Stretching | Active Laser | Control
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29 | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No